CLINICAL TRIAL: NCT06429865
Title: Safety and Effectiveness of Cytosponge in Surveillance After Endoscopic Submucosal Dissection for Esophageal Squamous Cell Carcinoma
Brief Title: Cytosponge in Surveillance After Endoscopic Submucosal Dissection for Esophageal Squamous Cell Carcinoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Tongliao City Hospital (Unknown); Ankang Central Hospital (Other); Yancheng First People's Hospital (Other); Lianshui County People's Hospital (Unknown); Nanchong Central Hospital (Other Government); Henan Provincial People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Zhongda Hospital (Other); Affiliated hospital of nanjing university hospital of Chinese medicine (Unknown)
Responsible Party: Principal Investigator, Wangluowei, PhD; MD； Chief Physician, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTSESD-20220509
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Cytosponge; Surveillance
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- esophageal squamous cell carcinoma group (Experimental): Participants were instructed to place the capsule near the root of the tongue and fold the string in their mouths, leaving approximately 20 cm of string outside, with a blue mark on the string right at the lips. The capsule was then swallowed with water, and the end of the string was held out of the mouth. Participants were then asked to slowly drink 150-200 mL of 50°C water in approximately 2 minutes to allow the capsule to dissolve so that the sponge mesh inside was released. The device was then slowly withdrawn up the esophagus by pulling the string. The retrieved and expanded cell collection material was put in preservative fluid (Froeasy Technology, Nanjing, China) and transferred to the cytology laboratory at room temperature.
  Interventions: Diagnostic Test: cytosponge

INTERVENTIONS:
Diagnostic Test: cytosponge — Use of cytosponge as a tool to patients who need surveillance after endoscopic submucosal dissection for esophageal squamous cell carcinoma

SUMMARY:
cytosponge has good diagnostic efficacy in the diagnosis of esophageal cancer, and is more safe, economic and comfortable. It is expected to replace gastroscope in the surveillance after endoscopic submucosal dissection to a certain extent. At present, there is no relevant research at home and abroad. This study plans to establish a large sample cohort based on the collaborative research network established earlier, prospectively include 1000 patients who received endoscopic submucosal dissection for esophageal squamous cell carcinoma and compare the effectiveness and safety of cytosponge and gastroscope in surveillance after endoscopic submucosal dissection for esophageal squamous cell carcinoma through self -comparison.

DETAILED DESCRIPTION:
Esophageal cancer is one of the common malignant tumors in the world. In 2020, the number of new cases of esophageal cancer in the world will reach 604000, and the number of deaths will reach 544000. As a high incidence area of esophageal cancer in China, esophageal squamous cell carcinoma (ESCC) is the most common, with about 324000 cases of morbidity and 301000 deaths each year, posing a serious threat to people's lives and health. With the continuous development of digestive endoscopy technology, endoscopic submucosal dissection (ESD) and other minimally invasive endoscopic techniques have become the first line of treatment for early esophageal cancer. However, studies have shown that there is a risk of local recurrence within one year after ESD for early esophageal cancer, with a recurrence rate of 0-17%. Therefore, surveillance detection after ESD has become an important link in the diagnosis and treatment of esophageal cancer.

At present, there is no uniform standard at home and abroad for surveillance after ESD for esophageal squamous cell carcinoma, no matter the frequency or method of surveillance. For example, the guidelines issued by Japan suggest that the surveillance should be conducted every 6 to 12 months after ESD, at least once a year. In the guidelines issued by the European Society of Gastroenterology, it is recommended to review endoscopy 3 to 6 months after ESD. If there is no recurrence, it can be changed to review endoscopy once a year. The Guidelines for the Diagnosis and Treatment of Esophageal Cancer issued by the National Health Commission in April 2022 suggests that patients should be rechecked 3 months, 6 months and 12 months after ESD, and if there is no recurrence, they should be rechecked once a year. Recheck once every three months within two years after surgery, once every six months within two to five years, and once every year after five years. Although the above guidelines and specific strategies for surveillance after esophageal cancer surgery have not yet been unified, the use of upper gastrointestinal endoscopy (hereinafter referred to as "gastroscope") as the main means of review and close surveillance are more consistent.

However, due to the invasiveness, cost and availability of gastroscope, frequent endoscopic surveillance of patients with esophageal cancer after ESD may bring significant economic and health burden to patients, and lead to a decline in patients' subjective surveillance enthusiasm. Therefore, it is of great significance to find a more safe, economical and comfortable surveillance method that is equivalent to the diagnostic performance of gastroscope for standardizing the surveillance after ESD for esophageal cancer.

cytosponge is a new non-invasive examination method, which can diagnose esophageal lesions by collecting esophageal cells and carrying out cytological examination and p53 staining. Its diagnostic efficacy for esophageal cancer has been confirmed in various studies at home and abroad. Esophageal cytology has been proved to have a good application prospect in the identification and screening of high-risk groups of esophageal cancer. In the 20th century, our country widely carried out esophageal mesh cytology for screening esophageal cancer in high incidence areas, but this method has low sensitivity (39%~47%), is easy to miss diagnosis, and has poor inspection comfort, and has been eliminated at present. The improved new esophageal cell collectors (such as CytospongeTM, EsophaCapTM, Shikang No. 1 TM, etc.) adopt the expanded sponge capsule design, which increases the contact area with esophageal mucosa, and has a higher success rate than the original dragnet cytology sampling. Cytological examination is relatively simple. Combining with the high-risk factor scoring scale can improve the screening effect and improve the positive rate and screening efficiency of surveillance endoscopic intensive examination. Foreign studies on Barrett's esophagus showed that the sensitivity of cytology combined with different biomarkers of the new cell collector of the esophagus was 73.3% - 93.1%, and the specificity was 92.4-95.7%; It can play a good risk stratification role in Barrett's esophageal related dysplasia and early esophageal adenocarcinoma (0% in low-risk group, 14% in medium risk group, and 87% in high-risk group). The diagnostic and management guidelines for Barrett's esophagus formulated by the British Gastroenterological Association and the American Gastroenterological Society both point out that: Cytosponge can be used as a screening method for Barrett's esophagus, and it is more in line with the principles of health economics. As early as 2010, a prospective cohort study in the UK showed that the sensitivity and specificity of cytosponges in diagnosing Barrett's esophagus with a circumference of 1cm or more were 73.3% and 93.8%, respectively. Similarly, a multicenter randomized controlled trial in the UK in recent years also confirmed the diagnostic efficacy of cellular sponge capsule in Barrett's esophagus. In addition, for areas with high incidence of ESCC, a study based on the Golestan cohort in Iran pointed out that the accuracy of cytological examination combined with p53 staining in detecting high-grade esophageal squamous hyperplasia could reach 100%. In a previous study conducted by our team, 1844 subjects from high-risk areas of ESCC were recruited, and the effectiveness, safety and comfort of the two in esophageal cancer screening were compared through cytosponge examination and gastroscopy. The results showed that the sensitivity and specificity of cellular sponge capsule in the diagnosis of high-grade esophageal lesions (including esophageal squamous cell carcinoma and high-grade intraepithelial neoplasia) were 90% and 93.7% respectively. However, no serious adverse events were recorded during cell collection, which fully demonstrates the feasibility and safety of AI helper cytosponge in community screening of ESCC.

To sum up, the cellular sponge capsule has good diagnostic efficacy in the diagnosis of esophageal cancer, and is more safe, economical and comfortable. It is expected to replace gastroscope in the surveillance after ESD to a certain extent. At present, there is no relevant research at home and abroad. This study plans to establish a large sample cohort based on the collaborative research network established earlier, prospectively include 1000 patients who received ESD resection treatment for early esophageal cancer and compare the effectiveness and safety of cytosponge and gastroscope in the surveillance of early esophageal cancer after ESD through self-comparison.

ELIGIBILITY:
Inclusion Criteria:

* (1) Sex unlimited, age 18-85; (2) The indication of ESD for early (superficial) esophageal squamous cell carcinoma conforms to the domestic and foreign guidelines; (3) The pathological stage of ESD was pT1a/pT1b.

Exclusion Criteria:

* (1) The pathological findings after ESD were HGIN; (2) Dysphagia (Stooler grade 2-4), inability to swallow cell sponge capsule successfully; (3) Postoperative pathological data were incomplete; (4) Have a history of cancer, early cancer, adenoma and other benign and malignant tumors of stomach and duodenum, combined with malignant tumors of other parts; (5) Previous esophageal or gastric surgery; (6) Esophagectomy, segmented endoscopic mucosal resection (EMR), multi ring mucosal resection (MBM) and other endoscopic non block resection techniques were used; (7) Those who have coagulation dysfunction or need to take anticoagulant and antiplatelet drugs continuously; (8) There are contraindications to gastroscopy and mucosal biopsy; (9) People with other serious diseases whose life expectancy is less than 5 years; (10) I refuse to cooperate with the research scheme and refuse to sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 60 minute
  Sensitivity and Specificity

CONTACTS AND LOCATIONS:
Overall Officials: Luowei Wang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No